CLINICAL TRIAL: NCT06749548
Title: A Comparison of Multidetector Computed Tomography and Transthoracic Echocardiography in the Diagnosis of Congenital Cyanotic Heart Diseases
Brief Title: A Comparison of Multidetector CT and TE in the Diagnosis of Congenital Cyanotic Heart Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/042
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Group 1 — the study is to emphasize the role of Computed Tomography Angiography (MDCTA) and Transthoracic Echocardiography (Echo) in the diagnosis of congenital cyanotic heart diseases.

SUMMARY:
Multi-detector computed tomography angiography (MDCTA) provides high-resolution images of the heart and its vasculature, allowing for accurate anatomical assessment, detection of complex cardiac morphology,

DETAILED DESCRIPTION:
evaluation of coronary artery anatomy, and identification of extracardiac anomalies including the coronaries, pulmonary arteries, aorta, and pulmonary or systemic veins, and it delineates vessel walls and also displays the airway, mediastinal abnormalities, and pulmonary parenchyma by using contrast media. This modality is particularly useful for evaluating complex cardiac anatomy and identifying potential surgical or interventional targets.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 and less than 65.
* having Congenital Cyanotic Heart Diseases

Exclusion Criteria:

* heart surgery
* other heart issues
* not consented

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the Aim is to compare the Multidetector CT and TE in the Diagnosis of Congenital Cyanotic Heart Diseases
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
Computed Tomgraphy Angiogrpahy | 12 Months
  All patients will undergo MDCT using a 128-slice scanner. A contrast agent will be administered to visualize the heart's vascular structures. Detailed images of the heart's chambers, major blood vessels, and defects will be acquired

CONTACTS AND LOCATIONS:
Locations (1):
- Timergara Teaching Hospital, Timergara District Dir Lower, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No